CLINICAL TRIAL: NCT05448755
Title: A Phase 2 Open Label Pilot Study to Evaluate the Safety and Efficacy of Subcutaneously Administered ELX-02 in Patients With Alport Syndrome With Col4A5 and Col4A3/4 Nonsense Mutation
Brief Title: A Study of ELX-02 in Patients With Alport Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EL-014
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-06

CONDITIONS: Alport Syndrome
Keywords: Aminoglycoside; Nonsense Mutation; Translational read through
MeSH Terms: conditions — Nephritis, Hereditary | interventions — ELX-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label study drug treatment (Experimental)
  Interventions: Drug: ELX-02

INTERVENTIONS:
Drug: ELX-02 — ELX-02 is a small molecule, new chemical entity being developed for the treatment of genetic diseases caused by nonsense mutations. ELX-02 is a eukaryotic ribosomal selective glycoside (ERSG).

SUMMARY:
This is a Phase 2 open label pilot study to evaluate the safety and efficacy of subcutaneously administered ELX-02 in patients with X-linked or autosomal recessive Alport Syndrome with Col4A5 and Col4A3/4 nonsense mutation.

In total, up to 8 participants, with a minimum of 3 adults, will be enrolled in the trial.

The study will be comprised of the following periods for each participant:

* a Screening period of up to 6 weeks (42 days)
* a total Treatment Period of 8 weeks (60 days)
* a safety/efficacy Follow-up Period of 12 weeks (90 days) after the last treatment The Treatment Period will be a treatment of ELX-02 0.75 mg/kg SC QD for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of X-linked or autosomal recessive Alport Syndrome with a documented nonsense mutation of Col4A5 in a male or nonsense mutation of Col4A3 or Col4A4 (male or female)
* The nonsense mutation should be UAG or UGA
* eGFR>60 ml/min/1.73 m2 (based on CKD-EPI for ages ≥18 and Schwartz formula for participants <18)
* Urinary protein based on two spot urine collections [urine protein/creatinine ratio (UPCR) ≥ 500 mg/g]
* Stable regimen of ACEi/ARB for at least 4 weeks before screening (unless there is a contraindication)

Exclusion Criteria:

* History of any organ transplantation
* Mutation consistent with autosomal dominant Alport Syndrome
* Liver disease characterized by cirrhosis or portal hypertension. Participants with alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or a total bilirubin 3.0 times the upper limit of normal (ULN) will be excluded
* History of congestive heart failure diagnosed clinically or with documented left ventricular ejection fraction (LVEF) ≤ 40%
* History of dialysis

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and characteristics of adverse events | From the time of first dosing through the end of the follow-up period, a total of 5 months

SECONDARY OUTCOMES:
Change in proteinuria | From screening assessment to end of study treatment and end of follow up period, two and five months respectively
Change in Col IV expression in renal biopsy | From biopsy collected at screening to the biopsy collected at the end of study treatment, a two months interval
Change in hematuria | From screening assessment to end of study treatment and end of follow up period, two and five months respectively

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - Monash Medical Center, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
- United Kingdom (2):
  - Royal Free Hospital, London
  - Great Ormond Street Hospital, London

REFERENCES:
- [Derived] Rheault MN. Treatment Approaches for Alport Syndrome. J Am Soc Nephrol. 2025 Sep 12;37(1):172-9. doi: 10.1681/ASN.0000000897. Online ahead of print. PMID 40938675
- See also: Eloxx Pharmaceuticals Website — http://www.eloxxpharma.com